CLINICAL TRIAL: NCT02410811
Title: Novel Cardiac Magnetic Resonance Imaging to Define a Unique Restrictive Cardiomyopathy in Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-4851
Record Dates: First submitted 2014-05-02; First posted 2015-04-08 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2019-06

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease (SCD); Cardiac Magnetic Resonance Imaging (CMR); Cardiomyopathy; Pulmonary Hypertension
MeSH Terms: conditions — Anemia, Sickle Cell; Cardiomyopathies; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, DNA, and urine specimens.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Age Stratum A: * Age 6 to 13.99 years
  * Cardiac magnetic resonance imaging (CMR)
  Interventions: Other: Cardiac magnetic resonance imaging (CMR)
- Age Stratum B: * Age 14 to 20.99 years
  * Detectible and quantifiable TRJV with reported value
  * Cardiac magnetic resonance imaging (CMR)
  Interventions: Other: Cardiac magnetic resonance imaging (CMR)
- Age Stratum C: * Age ≥21 years
  * Detectible and quantifiable TRJV with reported value
  * Cardiac magnetic resonance imaging (CMR)
  Interventions: Other: Cardiac magnetic resonance imaging (CMR)
- Age Stratum D: * Age ≥6 years.
  * Current use of disease-modifying therapy [hydroxyurea, chronic transfusions, or both (given concurrently, sequentially, or both)] that was initiated at <3 years of age, and for which there has been no interruption of therapy for >6 consecutive months since the initiation of disease-modifying therapy.
  * Cardiac magnetic resonance imaging (CMR)
  Interventions: Other: Cardiac magnetic resonance imaging (CMR)

INTERVENTIONS:
Other: Cardiac magnetic resonance imaging (CMR) — CMR is obtained on all participants in all arms/groups

SUMMARY:
The purpose of this study is to use cardiac magnetic resonance imaging (CMR) and echocardiographic tissue Doppler imaging to demonstrate a unique restrictive cardiomyopathy of sickle cell disease. The investigators will characterize its frequency and how it might change (e.g., presence/absence and severity) over a 2-year period.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) causes progressive cardiopulmonary morbidity, beginning in childhood, which can ultimately be fatal. As a group, cardiopulmonary complications, such as acute chest syndrome and sudden death, are now the most common causes of death in SCD, especially in adolescents and adults.

Patients with SCD have features of both an anemia-related, high cardiac output state and a restrictive cardiomyopathy (RCM). The investigators propose that this unique RCM is an overlooked and understudied complication of SCD. RCM could explain the modest increases in pulmonary artery pressure in patients with SCD, as measured by cardiac catheterization or estimated by tricuspid regurgitant jet velocity (TRJV), which has often been attributed to a primary pulmonary arterial hypertension (PAH). RCM could also be the cause of unexplained sudden cardiac death in SCD, which is a feature of other forms of RCM.

The investigators overarching hypothesis is that increased reactive oxygen species (ROS)-mediated angiotensin-1 receptor (AT1R)-TGFβ1 signaling is pro-fibrotic and, in combination with vaso-occlusive ischemia-reperfusion injury, results in an age-dependent, progressive RCM that can be detected by non-invasive cardiac imaging.

This pilot, longitudinal, observational study uses a novel, comprehensive, multimodal cardiac imaging strategy, combining cutting-edge cardiac magnetic resonance imaging (CMR) and echocardiographic tissue Doppler imaging (TDI), to demonstrate the unique RCM of SCD, characterizing its frequency and the temporal evolution over a 2-year period. The investigators will also correlate the RCM phenotype with biomarkers of ROS and renin angiotensin system (RAS)-TGFβ1 signaling.

This research could change the investigators understanding of how SCD affects the heart and lungs. The investigators propose studies that will change the current concept of primary pulmonary vasculopathy to a cardiomyopathy-centered model with secondary pulmonary vascular changes leading to sudden death. This translational pilot study will deliver a novel, clear, quantifiable CMR phenotype with established diagnostic performance that will be used in phase II/III clinical trials to test anti-fibrotic therapy to prevent or reverse SCD-related RCM.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell anemia (HbSS) or sickle-β°-thalassemia (HbSβ°) confirmed by hemoglobin separation and identification techniques
* Ability to cooperate with and undergo CMR without sedation or anesthesia.
* Ability to cooperate with and undergo echocardiogram
* Written informed consent in accordance with the institutional policies and federal guidelines must be provided by the participant (if ≥18 years of age) or parent or legally authorized guardian (if the participant is <18 years of age) Minor participants ≥11 years of age will be requested to provide assent

The following additional inclusion criterion applies to Age Stratum A:

Age 6 to 13.99 years

The following additional inclusion criteria apply to Age Stratum B:

* Age 14 to 20.99 years
* Detectible and quantifiable TRJV with reported value

The following additional inclusion criteria apply to Age Stratum C:

* Age ≥21 years
* Detectible and quantifiable TRJV with reported value

The following additional inclusion criteria apply to Stratum D:

* Age ≥6 years.
* Current use of disease-modifying therapy [hydroxyurea, chronic transfusions, or both (given concurrently, sequentially, or both)] that was initiated at <3 years of age, and for which there has been no interruption of therapy for >6 consecutive months since the initiation of disease-modifying therapy.

Exclusion Criteria:

* Any contraindication to MRI or physical or behavioral factor that could degrade the quality of MRI data or interfere with a participant's tolerance of the MRI, such as permanent or semi-permanent metallic implants, including pacemakers and defibrillators, or severe claustrophobia
* Known ventricular septal defect (VSD) documented in medical record
* Estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73 m2 (estimated by serum creatinine or cystatin-C)
* Pregnancy (documented by serum or urine pregnancy test)

The following additional inclusion criterion applies to strata A, B and C only:

- Current chronic transfusion therapy (defined as regular, approximately monthly, transfusions of packed red blood cells given for at least 6 consecutive months for the treatment of prevention of SCD-related complications with the plan to continue this therapy at the time of potential enrollment).

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Enrolling a maximum of 40 participants in the entire study across four age strata: A, 6 - 13.9 years; B, 14 - 20.9 years; C, 21 years and older; and D, 6 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-01-31; Primary Completion 2018-01-29 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles T Quinn, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati; Michael D Taylor, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Robert J Fleck, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati; Omar Y Niss, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Powell AW, Alsaied T, Niss O, Fleck RJ, Malik P, Quinn CT, Mays WA, Taylor MD, Chin C. Abnormal submaximal cardiopulmonary exercise parameters predict impaired peak exercise performance in sickle cell anemia patients. Pediatr Blood Cancer. 2019 Jun;66(6):e27703. doi: 10.1002/pbc.27703. Epub 2019 Mar 7. PMID 30848046
- [Result] Alsaied T, Niss O, Powell AW, Fleck RJ, Cnota JF, Chin C, Malik P, Quinn CT, Taylor MD. Diastolic dysfunction is associated with exercise impairment in patients with sickle cell anemia. Pediatr Blood Cancer. 2018 Aug;65(8):e27113. doi: 10.1002/pbc.27113. Epub 2018 May 21. PMID 29781568
- [Result] Niss O, Fleck R, Makue F, Alsaied T, Desai P, Towbin JA, Malik P, Taylor MD, Quinn CT. Association between diffuse myocardial fibrosis and diastolic dysfunction in sickle cell anemia. Blood. 2017 Jul 13;130(2):205-213. doi: 10.1182/blood-2017-02-767624. Epub 2017 May 15. PMID 28507082
- [Result] Niss O, Quinn CT, Lane A, Daily J, Khoury PR, Bakeer N, Kimball TR, Towbin JA, Malik P, Taylor MD. Cardiomyopathy With Restrictive Physiology in Sickle Cell Disease. JACC Cardiovasc Imaging. 2016 Mar;9(3):243-52. doi: 10.1016/j.jcmg.2015.05.013. Epub 2016 Feb 17. PMID 26897687
- [Derived] Niss O, Morin CE, Hashemi S, Alsaied T, Lang SM, Taylor MD, Tasset M, Malik P, Quinn CT. Longitudinal changes and predictors of cardiac extracellular volume fraction in sickle cell anemia. Blood Red Cells Iron. 2025 Dec;1(3):100031. doi: 10.1016/j.brci.2025.100031. Epub 2025 Nov 20. PMID 41312339

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum A (6-13.99 Years): * Age 6 to 13.99 years.
  * Sickle cell anemia or sickle-β0-thalassemia.
- Stratum B (14-20.99 Years): * Age 14 to 20.99 years.
  * Sickle cell anemia or sickle-β0-thalassemia.
  * Detectible and quantifiable tricuspid regurgitant jet velocity (TRJV).
- Stratum C (≥21 Years): * Age ≥21 years.
  * Sickle cell anemia or sickle-β0-thalassemia.
  * Detectible and quantifiable tricuspid regurgitant jet velocity (TRJV).
- Stratum D (Early Treatment): * Age ≥6 years.
  * Sickle cell anemia or sickle-β0-thalassemia.
  * Current use of disease-modifying therapy [hydroxyurea, chronic transfusions, or both (given concurrently, sequentially, or both)] that was initiated at <3 years of age, and for which there has been no interruption of therapy for >6 consecutive months since the initiation of disease-modifying therapy.
Period: Overall Study
Arm/Group | Stratum A (6-13.99 Years) | Stratum B (14-20.99 Years) | Stratum C (≥21 Years) | Stratum D (Early Treatment)
Started | 5 | 10 | 11 | 7
Completed | 5 | 10 | 10 | 7
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum A (6-13.99 Years) | Stratum B (14-20.99 Years) | Stratum C (≥21 Years) | Stratum D (Early Treatment) | Total
Number analyzed (Participants) | 5 | 10 | 11 | 7 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 6 | 0 | 5 | 16
  Between 18 and 65 years | 0 | 4 | 11 | 2 | 17
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.0 (9.2) | 18.0 (9.1) | 35.8 (13.1) | 13.4 (6.9) | 22.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8 | 4 | 20
  Male | 2 | 5 | 3 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 10 | 11 | 7 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 10 | 11 | 7 | 33
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 | 11 | 7 | 33
Sickle cell disease genotype [Count of Participants; unit: Participants]
  Homozygous sickle cell anemia (HbSS) | 4 | 10 | 11 | 7 | 32
  Sickle-β0-thalassemia (HbSβ0) | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency of the Diffuse Myocardial Fibrosis Phenotype
Description: The occurrence of an abnormally increased extracellular volume (ECV) measurement [i.e., the presence of the diffuse myocardial fibrosis phenotype] as assessed by cardiac magnetic resonance imaging (CMR) using T1 mapping before and after administration of gadolinium. Expressed as number of participants with the diffuse myocardial fibrosis phenotype in each stratum.
Time Frame: Assessed annually over a 2-year period (3 assessments over 2 years)
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum A (6-13.99 Years) | Stratum B (14-20.99 Years) | Stratum C (≥21 Years) | Stratum D (Early Treatment)
Number analyzed (Participants) | 5 | 10 | 10 | 7
Participants | 5 | 10 | 10 | 1

2. Other Pre Specified Outcome: Stability of the Diffuse Myocardial Fibrosis Phenotype Over Time
Description: The occurrence of a change [from the baseline assessment] in the classification [presence or absence] of the diffuse myocardial fibrosis phenotype, which is defined as an abnormally increased extracellular volume (ECV) measurement as assessed by cardiac magnetic resonance imaging (CMR) using T1 mapping before and after administration of gadolinium. Expressed as number of participants who had a change in classification of the diffuse myocardial fibrosis phenotype [e.g., presence to absence, or absence to presence] during the 2-year study in each stratum.
Time Frame: Assessed annually over a 2-year period (3 assessments over 2 years)
Population: Stratum D participants had a single CMR assessment only; no longitudinal data were collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum A (6-13.99 Years) | Stratum B (14-20.99 Years) | Stratum C (≥21 Years) | Stratum D (Early Treatment)
Number analyzed (Participants) | 5 | 10 | 10 | 0
Participants | 0 | 0 | 0 |

ADVERSE EVENTS:
Time Frame: AEs were collected for three, separate 30-day intervals over the entire study period of 2 years. Each 30-day interval was defined as starting with the study visit during which annual study activities were performed (e.g., cardiac magnetic resonance imaging [CMR]) and ending 30 days after that study visit. AEs were assessed as they occurred during each study visit, and AEs that occurred in the 30 days after each study visit were collected by scripted phone call from the study team.
Arm/Group | Stratum A (6-13.99 Years) | Stratum B (14-20.99 Years) | Stratum C (≥21 Years) | Stratum D (Early Treatment)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/10 | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/10 | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 3/10 | 1/10 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A (6-13.99 Years) (N=5) | Stratum B (14-20.99 Years) (N=10) | Stratum C (≥21 Years) (N=10) | Stratum D (Early Treatment) (N=7)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaso-occlusive pain episode (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — Sickle cell pain crisis

LIMITATIONS AND CAVEATS:
All participants in strata A, B and C had severe diffuse myocardial fibrosis. That is, all participants had the phenotype for which we assessed, so correlative studies (e.g., affected vs. non-affected) could not be performed. Therefore, we amended the protocol and opened an additional, fourth stratum (D) to study individuals who were previously not eligible for inclusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT02410811/Prot_SAP_000.pdf